CLINICAL TRIAL: NCT01153646
Title: A Pilot Study of Safety and Feasibility of T-Cell Immunotherapy Using Lentivirus Vector-Expressed RNAi in Autologous T-Cells of HIV-1 Infected Patients Who Have Failed Anti-Retroviral Therapy
Brief Title: Gene Transfer for HIV Using Autologous T Cells
Acronym: Gene Transfer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: John A. Zaia, MD, Principal Investigator Professor & Chair, Deptartment of Virology, Beckman Research Institute of City of Hope
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 03161; IND #14146 (Other: FDA)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: HIV-1 Infection
Keywords: HIV; Gene Transfer; T-Cell Immunotherapy; HIV-1 infected patients who have failed anti-retroviral therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort 1: 1x10e9 and Cohort 2: 1x10e10 T cells per infusion (Experimental): Group of patients receiving genetically modified T-cells
  Interventions: Genetic: pHIV7-shI-TAR-CCR5RZ treated CD4 cells

INTERVENTIONS:
Genetic: pHIV7-shI-TAR-CCR5RZ treated CD4 cells — Single dose administration x 3 of genetically modified T-cells given at 3 infusions at 6 week intervals.

SUMMARY:
This is a pilot study to determine the safety and feasibility of lentivirus-transduced T-cell immunotherapy in patients who have failed highly active anti-retrovirus therapy (HAART).

DETAILED DESCRIPTION:
Study Design This is a pilot study to determine the safety and feasibility of lentivirus-transduced T cell immunotherapy in patients who have failed highly active anti-retrovirus therapy (HAART) as defined by HIV levels or by intolerance to drug therapy. The lentivirus vector induces 3 forms of anti-HIV RNA: RNAi in the form of a short hairpin RNA (shRNA) targeted to an exon in HIV-1 tat/rev (shI), a decoy for HIV TAT-activated RNA (TAR), and a ribozyme that targets the host T cell CCR5 cytokine receptor (CCR5RZ). The vector is called rHIV7-shI-TAR-CCR5RZ and will be used in the transduction and expansion of autologous CD4-enriched T cells. Doses of 1 x 109 T cells will be given at 0, +6, and +12 weeks to the first cohort of 3 subjects. Following completion of this cohort, if no serious adverse events have occurred within 3 weeks of the last infusion, then the next cohort will receive 10 x 109 T cells at 0, +6, and +12 weeks using the same 8 week spacing between subjects.

Study Endpoints:

The primary endpoints of this pilot study are patient safety and study feasibility. Safety will be determined by clinical and laboratory observation and grading of adverse events, analysis of T cell repertoire clonality, and evaluation of HIV isolates for evidence of vector recombination. Feasibility will be determined by the ability to obtain suitable numbers of expanded T cells and expression of the RNA transgenes in these cells. The secondary endpoints are the duration of T cell circulation in blood post-infusion and the effect of the T cell infusion on CD4 count and on HIV load. Conventional CD4 counts and HIV RNA levels in blood will be determined at follow-up intervals.

Subject Eligibility and Number. Subjects must be HIV-1 infected adults ≥18 and ≤60 years of age who have been on HAART therapy for at least one year and have evidence of virologic failure defined by >5000 HIV RNA genome copies (gc) per mL in blood. Subjects must have a CD4 count of at least 200 CD4+ T cells/mL. This pilot study is expected to accrue five evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

Patient must:

* Be Age ≥ 18 years ≤ 60 years.
* Be HIV seropositive and have been treated with a potent antiretroviral chemotherapy regimen for at least one year and with an HIV plasma RNA >5000 gc/ml.
* Have available genotypic evidence of resistance and prior HAART modifications must have been consistent with current recommendations.
* Have a CD4 count >200 cells/mL and a CD4/CD8 ratio >0.2, with hemoglobin, WBC, and platelet count within 1.5x normal limits.
* Have a Karnofsky performance status >/= 70%.
* Have pretreatment SGOT, SGPT, and serum bilirubin <2.5 times the institutional upper limit of normal (ULN) with no extrinsic hepatobiliary disease and no HBV surface antigen and no hepatitis C virus antibody.
* Have PT/PTT <2 times the ULN.
* Have serum creatinine < 2 x ULN.
* Females Only: Must not be pregnant based on a pregnancy test within the past 7 days.
* Have CD4 counts are ≤ 200, is the patient on a prophylactic regimen for pneumocystis pneumonia or have they agreed to begin such treatment.
* Agree to use effective birth control to prevent pregnancy.
* Voluntarily consent and comply with the treatment and required tests.

Exclusion Criteria:

Patients are ineligible if:

* The patient has an active bacterial or fungal infection.
* The patient has been successfully treated AIDS related opportunistic infections within the past year.
* The patient has active CMV retinitis or other active CMV-related organ dysfunction (excluding completely treated CMV infections).
* The patient has evidence of clinically significant neuropathy.
* The patient has had a relapse of pneumocystis carinii pneumonia within the past year.
* The patient has intractable and severe diarrhea as defined as >1500 cc diarrheal fluid per day or diarrhea causing persistent severe electrolyte abnormalities or hypoalbuminemia.
* The patient has other AIDS-related syndromes, infections or other illness that would preclude autologous HCT as determined by the Principle Investigator.
* The patient has taken any immunosuppressive medications in the past 30 days.
* Has any prior malignancy, except those treated with curative intent that are five years from treatment, cervical and anal squamous cell cancers and superficial basal cell and squamous cell cancers of the skin.
* The patient has auto-antibodies.
* The patient has had a leukapheresis in the past 3 months.
* The patient has a known allergy to human serum albumin, Dextran 40 or DMSO.
* The patient has ever been on a gene therapy trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Patient Safety | Every 3 months for the first year, then twice yearly until year 5, and then yearly until year 15 after treatment
  Patient safety will be determined by clinical and laboratory observation and grading of adverse events using the CTCAE v.3. Assays: analysis of T cell repertoire clonality, and evaluation of HIV isolates for evidence of vector recombination.
Feasibility | Every 3 months for the first year, then twice yearly until year 5, and then yearly until year 15 after treatment
  Feasibility will be determined by the ability to obtain suitable numbers of expanded T cells and expression of the RNA transgenes in these cells. The secondary endpoints are the duration of T cell circulation in blood post-infusion and the effect of the T cell infusion on CD4 count and on HIV load. Conventional CD4 counts and HIV RNA levels in blood will be determined at follow-up intervals.

SECONDARY OUTCOMES:
Genetic marking in peripheral blood using vector-specific PCR assay. | During time of follow-up years 0-2

CONTACTS AND LOCATIONS:
Overall Officials: John A. Zaia, MD, Principal Investigator — Beckman Research Institute of City of Hope
Locations (1):
- Beckman Research Institute of City of Hope, Duarte, California, United States

REFERENCES:
- [Background] Levine BL, Bernstein WB, Aronson NE, Schlienger K, Cotte J, Perfetto S, Humphries MJ, Ratto-Kim S, Birx DL, Steffens C, Landay A, Carroll RG, June CH. Adoptive transfer of costimulated CD4+ T cells induces expansion of peripheral T cells and decreased CCR5 expression in HIV infection. Nat Med. 2002 Jan;8(1):47-53. doi: 10.1038/nm0102-47. PMID 11786906
- [Background] Sarver N, Cantin EM, Chang PS, Zaia JA, Ladne PA, Stephens DA, Rossi JJ. Ribozymes as potential anti-HIV-1 therapeutic agents. Science. 1990 Mar 9;247(4947):1222-5. doi: 10.1126/science.2107573.
- [Background] Bai J, Gorantla S, Banda N, Cagnon L, Rossi J, Akkina R. Characterization of anti-CCR5 ribozyme-transduced CD34+ hematopoietic progenitor cells in vitro and in a SCID-hu mouse model in vivo. Mol Ther. 2000 Mar;1(3):244-54. doi: 10.1006/mthe.2000.0038. PMID 10933940
- [Background] Bauer G, Valdez P, Kearns K, Bahner I, Wen SF, Zaia JA, Kohn DB. Inhibition of human immunodeficiency virus-1 (HIV-1) replication after transduction of granulocyte colony-stimulating factor-mobilized CD34+ cells from HIV-1-infected donors using retroviral vectors containing anti-HIV-1 genes. Blood. 1997 Apr 1;89(7):2259-67. PMID 9116267
- [Background] Lee NS, Dohjima T, Bauer G, Li H, Li MJ, Ehsani A, Salvaterra P, Rossi J. Expression of small interfering RNAs targeted against HIV-1 rev transcripts in human cells. Nat Biotechnol. 2002 May;20(5):500-5. doi: 10.1038/nbt0502-500. PMID 11981565
- [Background] Li MJ, Bauer G, Michienzi A, Yee JK, Lee NS, Kim J, Li S, Castanotto D, Zaia J, Rossi JJ. Inhibition of HIV-1 infection by lentiviral vectors expressing Pol III-promoted anti-HIV RNAs. Mol Ther. 2003 Aug;8(2):196-206. doi: 10.1016/s1525-0016(03)00165-5. PMID 12907142
- [Background] Li MJ, Kim J, Li S, Zaia J, Yee JK, Anderson J, Akkina R, Rossi JJ. Long-term inhibition of HIV-1 infection in primary hematopoietic cells by lentiviral vector delivery of a triple combination of anti-HIV shRNA, anti-CCR5 ribozyme, and a nucleolar-localizing TAR decoy. Mol Ther. 2005 Nov;12(5):900-9. doi: 10.1016/j.ymthe.2005.07.524. Epub 2005 Aug 22. PMID 16115802